CLINICAL TRIAL: NCT06793449
Title: A Prospective, Non-inferiority Study Comparing VRD±D Followed by BCMA CAR-T Cell Therapy Versus VRD±D Followed by Autologous Hematopoietic Stem Cell Transplantation in Transplant-eligible Patients With Newly-diagnosed Multiple Myeloma
Brief Title: BCMA CAR-T Versus ASCT in Transplant-eligible Patients With Multiple Myeloma
Acronym: CAREMM-006
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024104
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASCT (Active Comparator): Patients will receive 3-4 cycles induction treatment, and high-dose melphalan conditioning, followed by autologous transplantation.Three months post-transplant, patients will undergo 2-3 cycles of consolidation therapy, followed by maintenance therapy for ≥2 years or until disease progression, death, intolerance, withdrawal for other reasons, or the study's termination/completion.
  Interventions: Biological: ASCT
- BCMA CAR-T (Experimental): Patients will receives 3-4 cycles of induction therapy, 2-3 cycles of consolidation treatment, followed by Fc-based conditioning and CAR-T cell infusion. One month after CAR-T cell therapy, patients will begin maintenance therapy for ≥2 years or until disease progression, death, intolerance, withdrawal for other reasons, or the study's termination/completion.
  Interventions: Biological: anti-BCMA CAR-T

INTERVENTIONS:
Biological: anti-BCMA CAR-T — Autologous BCMA-directed CAR-T cells, infusion intravenously at a target dose of 2.0-4.0 x 10^6 anti-BCMA CAR+T cells/kg.
  Arms: BCMA CAR-T
Biological: ASCT — Autologous stem cell infusion
  Arms: ASCT

SUMMARY:
This is a prospective, non-inferiority study comparing VRD±D followed by BCMA CAR-T cell therapy versus VRD±D followed by autologous hematopoietic stem cell transplantation in the treatment of newly diagnosed multiple myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be informed and voluntarily sign the Informed Consent Form (ICF).
2. Age between 18 and 70 years (inclusive).
3. Have measurable disease meeting at least one of the following criteria: Serum M-protein ≥1 g/dL (>10 g/L) as detected by serum protein electrophoresis (SPEP), or quantifiable IgA or IgD levels for IgA or IgD-type myeloma; Urine M-protein ≥200 mg/24 hours; In cases where serum and urine M-protein do not meet the above thresholds, an abnormal free light chain (FLC) ratio (normal range: 0.26 to 1.65) and involved serum FLC ≥100 mg/L.
4. Confirmed expression of the BCMA target antigen on MM cells by flow cytometry or bone marrow immunohistochemistry.
5. Assessed by the investigator as transplant-eligible.

Exclusion Criteria:

1. Primary plasma cell leukemia.
2. Concurrent amyloidosis.
3. Involvement of the central nervous system (CNS).
4. Previous treatment with BCMA-targeted therapy or CAR-T cell therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Persistent MRD-negative rate | Up to 2 year
  achieving MRD-negative, as determined by NGS/NGF
Progression free survival (PFS) | Up to 5 year
  Progression free survival is defined as the time from the date of diagnosis to the date of first documented PD, as defined in the IMWG criteria, or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Complete response rate (CRR) | within 1 week after induction therapy, 1 month after the CAR-T cell infusion or ASCT, within 1 week after consolidation therapy
  CR or better is defined as percentage of participants who achieve a CR response or Stringent Complete Response (sCR) response accoording to the IMWG criteria
Duration of Remission(DOR) | Up to 5 year
  Duration from the first evaluation of at least partial remission (PR) to the onset of disease progression or death due to disease progression (whichever occurs first)
Overall Survival (OS) | Up to 5 year
  Overall survival is measured from the date of diagnosis to the date of the participant's death.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: No